CLINICAL TRIAL: NCT04274010
Title: PANenteric Crohn's Capsule Versus Ileo-Colonoscopy and Scan Study
Acronym: PAN-ICS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to meet recruitment target due to multitude of factors (strict eligibility criteria and lack of clinician and participant engagement)
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Collaborators: County Durham and Darlington NHS Foundation Trust (Other Government); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Newcastle University (Other); Durham University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 275854
Record Dates: First submitted 2020-01-22; First posted 2020-02-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Crohn Disease
Keywords: capsule endoscopy; ileocolonoscopy; magnetic resonance enterography
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crohn's capsule (Other): Single-arm non-randomised study, all participants will undergo MRE, ileo-colonoscopy and Crohn's capsule.
  Interventions: Diagnostic Test: PillCamTM Crohn's capsule; Diagnostic Test: Magnetic resonance enterography; Procedure: Ileo-colonoscopy

INTERVENTIONS:
Diagnostic Test: PillCamTM Crohn's capsule — Capsule endoscopy for small and large bowel to assess Crohn's disease activity.
Diagnostic Test: Magnetic resonance enterography — MRI scan of small bowel to assess small bowel Crohn's disease activity.
Procedure: Ileo-colonoscopy — Endoscopic procedure to assess Crohn's disease activity in colon and terminal ileum.

SUMMARY:
Crohn's disease (CD) is a lifelong condition affecting the small and/or large bowel, causing diarrhoea, abdominal pain and weight loss. Patients with CD receive two tests to assess if the patients' CD is active, namely ileo-colonoscopy (camera examination of the large bowel, IC) and a scan of the small bowel (MRE). Together, these tests help determine if the patients' symptoms are due to CD, which is important as the medication to heal the bowel is strong. But, these investigations are uncomfortable, embarrassing, time-consuming and involve hospital visits to two separate departments.

A new test involves swallowing a miniature camera, the size of a large vitamin pill (PillCam™ Crohn's (PCC)) that video-records the lining of the small and large bowel. Images are sent to a recorder worn over the tummy. The investigators aim to find out if the PCC capsule delivers a single test that is comparable to current tests (IC+MRE) for patients with CD.

125 patients with CD referred for IC+MRE will be recruited from 3 NHS hospitals. Each patient will undergo all three tests (IC+MRE and PCC). As there is a small risk of the capsule getting stuck (up to 3 in 100 patients), all patients will have a "dummy" capsule to check that the "real" capsule can travel safely through the bowel. If successful (checked with a handheld scanner and CT scan if required), patients proceed to PCC. Patients will receive bowel preparation (a drink to clean the bowel) prior to IC and PCC.

The investigators will compare the findings of all three tests. The investigators will interview patients to find out their experiences to inform the way the test is introduced into practice. When consulted, local patients with CD felt the research question is extremely important and all preferred having one non-invasive test over two invasive and uncomfortable tests.

DETAILED DESCRIPTION:
Purpose and design

Aims:

To determine if the PillCam™ Crohn's capsule (PCC) performs similarly to ileo-colonoscopy (IC) and magnetic resonance enterography (MRE) when assessing patients with an established diagnosis of Crohn's disease (CD).

Objectives:

Primary objective: To assess the number of positive results showing active disease which are detected ("positive yields") by PCC compared to IC and MRE in patients with an established diagnosis of CD.

Secondary objectives will focus on other performance characteristics of PCC in assessing CD and include the following:

* To investigate the association between the different scoring systems (MEGS, MaRIA, SES-CD, Lewis, CECDAIic) for severity of bowel inflammation for each test.
* To see if the clinical findings seen on PCC matches the clinical severity as graded by patients based on the Harvey-Bradshaw Index and patients' quality of life from the short IBD-Q.
* To assess the patient experience of each test in a smaller group of patients.

This study is a three-centre prospective non-randomised study held across three NHS hospital sites. The investigators will be recruiting 125 patients who have been referred for IC and MRE as part of standard NHS care to assess their CD. As part of this study, all patients will undergo the investigations as part of their routine care plus PCC so overall, the participants will undergo all three investigations, namely IC, MRE and PCC.

The three sites in this study are:

* South Tyneside District Hospital (STDH), South Tyneside and Sunderland NHS Foundation Trust (STSFT)
* Royal Hallamshire Hospital (RHH), Sheffield Teaching Hospitals NHS Foundation Trust (STH)
* Darlington Memorial Hospital (DMH), County Durham and Darlington NHS Foundation Trust (CDDFT) (not capsule endoscopy delivery site in delivering routine care)

DMH does not routinely deliver care for capsule endoscopy. Patients recruited from DMH will be referred to STDH for patency ("dummy") capsule and PCC. Whenever possible, the research team at STDH will perform both "dummy" capsule and PCC examinations in DMH to avoid patients travelling.

Recruitment

Study design and methodology:

Suitable patient candidates for the study will be identified in a gastroenterology clinic or an inflammatory bowel disease meeting. These patients will have been referred for both MRE and IC as part of their standard care. The clinician responsible for the patient's care will explore the patient's interest in participating in the study. Verbal consent to allow the research team to approach these patients will be gained by their responsible clinician either in clinic or via telephone.

These patients will be signposted to a research nurse or a clinical research doctor involved in the study at each hospital site. The research nurse and clinical research doctor would be authorised on the delegation log. The patient will be provided with a patient information sheet on the study and a patient information leaflet on the capsule procedures ("dummy" capsule and PCC) in clinic by either the patient's usual clinician or the research nurse. Alternatively, these documents could be sent to the patient in the post by the research team. The patient will also be given adequate time to consider participating in the study and be given an opportunity to ask questions about the study and about both the "dummy" capsule and PCC.

Following this, a patient may be approached or contacted by the patient's usual clinician (who will be authorised on the delegation log) or a member of the research team to discuss the study. A member of the research team at each hospital site will gain written consent from the patient to participate in the study. In addition to study participation consent, another form of written consent will be obtained for procedures such as IC (as part of standard care) and the "dummy" capsule and PCC (as part of research protocol). The consent forms used for the procedures are standard NHS consent forms used nationally. Specific consent will also be gained from the patient so that the investigators can inform the patient's General Practitioner of study participation.

All the study procedures and tests remain the same across all 3 hospital sites. Nevertheless, as CDDFT is not a hospital site which provides a capsule endoscopy service, suitable members of the research team who are trained in capsule endoscopy from STSFT will travel to CDDFT to gain consent from the participants for the "dummy" capsule and PCC, administer these and follow-up the participants' progress.

Once a patient has been consented, the patient will first undergo the MRE. This is important as the participant cannot have the scan if there is a retained capsule. The research team will coordinate patient appointments with the radiology and endoscopy department to ensure that the participant's MRE appointment occurs prior to the "dummy" capsule and PCC appointment.

All MRE results will be reviewed by the research team before the participants are given the "dummy" capsule. The participant proceeds to this unless the MRE shows a long fixed segment of small bowel narrowing (stricture) which is more than 30cm. In this case, the particular patient will be excluded from the study due to the risk of the capsule getting stuck within the bowel (capsule retention).

Within the 2 weeks following the MRE, the participant will attend the participant's local hospital site to have the "dummy" capsule. The participant does not need to drink bowel preparation (a drink to clean the bowel) for this. The participant will be supervised by a member of the research team while swallowing the "dummy" capsule at approximately 0800 hours. At approximately 1400 hours the following day, the participant will attend the hospital to assess the location of the "dummy" capsule. This involves using a handheld scanner. The investigators will not be able to use the handheld scanner on some patients who have a cardiac pacemaker or implanted cardiac defibrillator. These patients will have to undergo a limited CT scan to look for the location of the "dummy" capsule as recommended by the Sheffield Hospitals Trust. The limited CT scan will also be used if the handheld scanner is not available or if the scanner cannot detect the location of the "dummy" capsule.

If the participant pass the "dummy" capsule safely, the participant will proceed to PCC (and IC on the same day if possible) which will be scheduled as a separate appointment, usually within 3-5 working days. The patients who are found to have capsule retention will not be able to participate in the study. However, an appointment will be arranged to undergo IC as this was organised from the patients' recent clinic appointment. A retained "dummy" capsule will eventually dissolve itself in 72 hours and pass safely.

Before attending the appointment for PCC and IC, the participant will have to take bowel preparation the evening before. The participant may require additional bowel preparation and another appointment if IC cannot be performed on the same day as PCC. To avoid the need for bowel preparation to be taken twice, the research team will endeavour to ensure the appointments for PCC and IC coincide. The investigators acknowledge that this may not be feasible for all patients and appointments will be made at the convenience of patients.

Participants will be scheduled to arrive at the endoscopy department early in the morning (approximately 0730 hours). The participant will be supervised while swallowing the PCC to allow enough time for the capsule to pass. This gives the greatest chance of the participant being able to have the IC the same day. The progress of the capsule is monitored through the day. In a small number of patients who are unable to swallow the PCC or where it is delayed in travelling from the stomach into the small bowel, these patients will have a short camera test procedure (gastroscopy) to place the PCC in the small bowel. This is standard clinical practice under these circumstances and will be carried out after these patients have given additional consent. When the PCC is confirmed to have left the body, the participant proceeds to IC in the afternoon (approximately 1500 hours). Following this, the participant is discharged from hospital.

Anticipated situations where this may not occur include an incomplete capsule recording by the time of the participant's IC appointment later in the afternoon. If so, the recording of PCC is allowed to continue and the participant will be given the option of undergoing IC that afternoon (in which case the capsule would be encountered by the clinician performing the IC) or coming back on a different day (after further bowel preparation), within 2 weeks, for their IC.

The investigators would allow a 4-week period for participants to have all the investigations (MRE, "dummy" capsule, PCC and IC). Results from the MRE, PCC and IC will be recorded. Information about the participant's Crohn's disease, medication, recent blood or stool tests will be recorded. Participants would also be asked to complete a short quality of life questionnaire. All patients will have follow-up until all investigations are complete. Additionally, passage of the actual capsule (PCC) from the bowel will be confirmed with patients. If a patient is uncertain if it has passed, an X-ray of the abdomen will be arranged 2 weeks later at the patient's local hospital site.

A smaller group of 10-15 patients will be asked to attend an interview to evaluate the patients' experience relating to the PCC to see if this could be introduced into routine clinical care. At least 3 from each of the 3 sites will be selected. One-to-one interviews will be conducted and recorded on telephone by an experienced researcher (Dr Close). Interview schedules will be developed in collaboration with a patient group and interviews will be held at a time convenient to patients, between 1-6 weeks following the end of the patients' various investigations. The analysis will focus on how acceptable is the new test compared to usual care and patient views about its place in disease monitoring and management. Initial analysis will be conducted by Dr Close and the patient group will be consulted about the interpretation of findings.

As patients would have multiple hospital visits for IC and MRE as part of routine care, the investigators would attempt to minimise the number of additional hospital visits related to study consent, "dummy" capsule administration and follow-up. All patients are entitled to claim up to £25 to cover for any additional research-related hospital visits. This will be organised via the research nurse at each local hospital site.

Study calibration:

This study is designed in a way that the investigation and management pathway is reliable and can be readily applied to real-world routine practice. As such, interpreting and reporting scans and procedures will occur across all 3 hospital sites. Everyone involved in reporting these will have prior training to standardise report findings. For every patient's set of investigations, a clinician who reports a particular test for that patient will not have access or be made aware of the results of that same patient's other test results. This is to prevent any bias effect on all the report findings.

The approach to each investigation is described below:

* MRE: All MRE will be read locally. On top of standard reporting, all radiologists will be given training on how to calculate disease severity scores for the small bowel.
* PCC: All PCC will be read locally. Examinations performed at DMH will be read by someone at STDH. The data recorder will be securely transported between these 2 hospital sites. The data is encrypted and only accessible with specific reporting software. All readers will be experienced capsule endoscopy readers (reporting >75 capsule endoscopies per year). The capsule endoscopy readers will also have completed online learning provided by Medtronic (company that manufactures and provides PCC) and be given training on how to calculate disease severity scores when reporting.
* IC: All IC will be performed locally. Clinicians performing this procedure will be asked to report the IC by a standardised scoring system which details disease severity in the large bowel. Every effort will be made to access the last part of the small bowel (terminal ileum) to complete assessment but this may not sometimes be possible if patients have an inflamed bowel lining. These will be recorded. Tiny samples (biopsies) may be taken from the lining of the bowel if deemed necessary by the clinician performing the procedure.

As mentioned above, the clinicians reading PCC will be different from the clinicians performing IC. All clinicians will only have access to the results of the patient's investigation that the clinician is involved in reporting and not the other investigations.

Study information gathering:

The following information will be collected and recorded onto a paper case report form and then uploaded onto a secure online database (REDCap):

* Age
* Gender
* Reason for CD assessment
* Current Montreal-Paris classification of CD
* Current medication for CD
* Blood tests within 8 weeks prior to study entry: full blood count, urea & electrolytes, CRP, albumin
* Stool tests (faecal calprotectin) within 8 weeks prior to study entry
* Harvey-Bradshaw Index (HBI)
* Short IBDQ (IBD patient quality of life questionnaire)
* MRE results and disease severity scores
* IC results, biopsy results if applicable and disease severity score
* PCC results and disease severity scores

No follow-up (beyond confirmation of the passage of the PCC) is required for the study except for a subset of 10-15 patients recruited for interviews as stated above in "Study design and methodology". The duration of patient involvement in the study is from patient consent up to 4 weeks after the last investigation (MRE, IC or PCC). This is to allow time for the investigations to be carried out, reported, repeated if required and for data collection.

Results from IC and MRE will be managed in keeping with standard care. It is possible that subtle and abnormal small bowel findings are picked up by PCC that are not picked up by MRE. Results from PCC will be reviewed by the Principal Investigator of each hospital site and where the results differ from IC and MRE, this will be passed on to the patient's usual responsible doctor for further action if necessary.

Consent

Patients will be allowed adequate time to consider study participation. The patients will also be offered the opportunity to ask any questions. Written consent will be sought after a full explanation has been given by a fully-trained member of the research team. Additional written consent will be sought during the same session for all 3 procedures i.e. the "dummy" capsule, PCC and IC. A small proportion of patients who are selected for the telephone interview will have to sign a separate consent form for this purpose.

As participation in this study will require potentially one or more additional visits for the "dummy" capsule, or a further appointment for either PCC or IC if these cannot be performed on the same day, patients will be informed of this upon study participation. Additionally, the patients will be made aware that they may need to take bowel preparation twice. Participants will be reimbursed for research-related travel costs up to £25. This can be arranged via the participants' local hospital research team.

The patients will reserve the right to refuse to participate or withdraw at any time without affecting subsequent care. Any information collected up to that point will be recorded, unless participants specifically request that the investigators destroy any information collected.

Risks, burdens and benefits

Patients with CD often require two tests to assess if their CD is active, namely IC and MRE. These tests help determine if their symptoms are due to CD, which is important as medications to control the disease and heal the bowel lining are strong and expensive. However, these tests are uncomfortable, embarrassing, time-consuming and involve hospital visits to two separate departments.

The new test (PCC) involves swallowing a miniature camera, the size of a large vitamin pill that video-records the lining of the small and large bowel. Images are sent to a recorder worn over the tummy. This proposed study includes PCC, IC and MRE, therefore all findings within the entire small bowel and colon are compared between these tests. The investigators aim to assess how PCC performs in comparison to IC+MRE when assessing the severity of a patient's CD activity. There have not been prior studies comparing PCC to a combined set of IC+MRE which is more reflective of current standards of care. The outcome of this study will therefore be more readily applicable to standard practice.

If PCC delivers a single test that is comparable to current tests (IC+MRE) for patients with CD, then not only does it address issues patients have over having an invasive and potentially uncomfortable test (IC), but it also reduces the number of tests that patients need to have and visits to different hospital departments. It means fewer test results to wait for and lesser delay in treatment decisions, on top of saving cost and relieving huge pressure on radiology departments and endoscopy units which are trying to meet all demands on their service.

Anticipated adverse events from this study could be related to either procedure (PCC or IC).

Adverse events (AE):

1. Retained "dummy" capsule or retained PCC
2. Bleeding or perforation (damage or puncture to the bowel lining) related to IC

Serious adverse events (SAE):

1. Unplanned admission to hospital due to retained "dummy" capsule or PCC
2. Camera test procedure (endoscopy) or an operation to remove the retained "dummy" capsule or PCC
3. Unplanned admission to hospital following IC or MRE which are directly related to the investigations

A retained capsule is defined as the presence of capsule two weeks after first swallowing it and where its passage from the bowel has not been detected. This can also happen if a patient starts developing symptoms strongly suggestive of a blockage within the bowel after swallowing the capsule. Side effects from bowel preparation such as nausea, vomiting, abdominal pain and bloating are not included as an adverse event. Each AE or SAE will be recorded in an adverse event form and the sponsor, trials steering committee and independent data monitoring committee will be notified.

Risks of retained capsule will be minimised by reviewing the MRE results to ensure there are no strictures before they are given to patients. Patients will be given a "dummy" capsule which can self-dissolve and pass spontaneously even if it is stuck before being given the actual PCC. This would help exclude the group of patients who have strictures which are not visible on MRE.

The IC will be performed by fully qualified endoscopists so the risks of bleeding or perforation are very small (1 in 1000 chance).

The radiation exposure that the patient might receive over the course of the study (assuming 2 abdominal X-rays and 2 limited CT scans) could very slightly increase the risk of getting cancer. The normal risk of developing cancer at some point is 50% i.e. 1 in 2. The patient's total risk, including the risks from the scans involved in the patient's participation in the trial, would become 50.05% i.e. an increase of 0.05%. This increase in risk is considered to be low.

Confidentiality

The Caldicott Principles and General Protection Data Regulation (GPDR) will be fully adhered to when dealing with patient identifiable data. The Chief Investigators will preserve the confidentiality of participants taking part in the study. The data will be held at the site in accordance with local Trust policies and will be destroyed following the study has closed in accordance with local Research and Development protocols.

Patients will be informed upon study consent that relevant sections of their hospital notes, endoscopy records, laboratory results and biopsy samples will be accessed by a member of the research team. Results of PCC will not be anonymised to allow the investigators to match the participant's findings to the IC and MRE. Any information collected and uploaded onto the secure online database will be allocated a unique study ID for each patient with no identifiable information. No patient identifiable information will be passed outside of the participating Trusts. Any results published as part of this study will be anonymised.

All members of the research team will be trained in Good Clinical Practice in Research which is in line with the National Institute for Health Research policy. All those dealing with data will receive GDPR training and the study will be registered with the Caldicott Guardian at each hospital site.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Established diagnosis of Crohn's disease
* Patients who have been referred for IC and MRE for CD assessment as deemed appropriate by referring clinician as part of standard care

Exclusion Criteria:

* Indeterminate colitis or ulcerative colitis
* Stricturing disease - history consistent with obstruction e.g. nausea, vomiting, abdominal pain, bloating after meals or stricture seen on previous imaging
* Enteric fistulating disease based on clinical examination or previous imaging (perianal fistulae alone is allowed in the absence of anal strictures)
* Previous small bowel or colonic resection within 12 months
* Known or suspected bowel dysmotility
* Previous pelvic radiotherapy
* Insulin-treated diabetes mellitus
* Pregnancy
* Recent non-steroidal agent use within 4 weeks of study entry (excluding aspirin <150mg per day)
* Contraindications to MRE, IC or capsule endoscopy
* Contraindications to taking bowel preparation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Positive yields in Crohn's capsule vs ileo-colonoscopy and magnetic resonance enterography. | 4-6 weeks
  To assess the rate of macroscopically detectable disease or "positive yields" by the PillCamTM Crohn's capsule compared to ileo-colonoscopy and magnetic resonance enterography in patients with an established diagnosis of Crohn's disease.

SECONDARY OUTCOMES:
Correlation between small bowel scoring systems. | 4-6 weeks
  To determine the correlation of small bowel scoring systems i.e. between the Lewis score for PillCamTM Crohn's capsule and the small bowel score of Magnetic Resonance Enterography Global Score (MEGS) and the small bowel Magnetic Resonance Index of Activity (MaRIA) score for MRE.
Correlation between colonic scoring systems. | 4-6 weeks
  To determine the correlation of colonic scoring systems i.e. between the colonic score of Capsule Endoscopy Crohn's Disease Activity Index for the Small Bowel and Colon (CECDAIic) for PillCamTM Crohn's capsule and the Simple Endoscopic Score for Crohn's Disease (SES-CD) for ileo-colonoscopy.
Positive diagnostic yield of Crohn's capsule with clinical severity of Crohn's disease. | 4-6 weeks
  To compare the positive diagnostic yield of PillCamTM Crohn's capsule with clinical severity based on the Harvey-Bradshaw Index.
Positive diagnostic yield of Crohn's capsule with patient quality of life. | 4-6 weeks
  To compare the positive diagnostic yield of PillCamTM Crohn's capsule with patient quality of life based on the short Inflammatory Bowel Disease-Questionnaire (IBD-Q) score.
Patient experience in each modality. | 4-6 weeks
  Qualitative assessment via telephone interview to evaluate a subset of patients based on their experience of undergoing PillCamTM Crohn's capsule endoscopy, MRE and ileo-colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Panter, Study Chair — South Tyneside and Sunderland NHS Foundation Trust
Locations (1):
- South Tyneside District Hospital, South Shields, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No